CLINICAL TRIAL: NCT02697474
Title: Persistence of Anti-Hep B Antibodies at 9 to 10 Years of Age in Subjects Having Received Hep B Vaccine at Birth and a DTaP-IPV-Hep B-PRP-T Hexavalent Vaccine at 2, 4 and 6 Months of Age, and Evaluation of Their Immune Memory Following a Challenge Re-vaccination With a Stand Alone Hep B Vaccine
Brief Title: Anti-Hep B Antibodies at Age 9 to 10 Years After Hep B Vaccine at Birth and DTaP-IPV-Hep B-PRP-T Hexavalent Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L49; U1111-1161-2421 (Other: WHO)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; DTaP-IPV-Hep B-PRP-T Hexavalent Vaccine; Euvax-B®; Hexaxim®; Infanrix® hexa
MeSH Terms: conditions — Hepatitis B | interventions — Euvax-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hexaxim® Group (Experimental): Subjects that received Hexaxim® in Study A3L12
  Interventions: Biological: Euvax B®: Hepatitis B vaccine
- Infanrix® hexa Group (Experimental): Subjects that received Infanrix® hexa in Study A3L12
  Interventions: Biological: Euvax B®: Hepatitis B vaccine

INTERVENTIONS:
Biological: Euvax B®: Hepatitis B vaccine — 0.5 mL, Intramuscular
  Other Names: Euvax B®
  Arms: Hexaxim® Group
Biological: Euvax B®: Hepatitis B vaccine — 0.5 mL, Intramuscular
  Other Names: Euvax B®
  Arms: Infanrix® hexa Group

SUMMARY:
The aim of the study is to assess the persistence of anti-Hep B antibody at 9 to 10 years of age after the last priming dose in subjects who completed study A3L12 (NCT00401531), and also evaluate the immune response against hepatitis B one month after vaccination (challenge vaccination) with a stand alone monovalent hepatitis B vaccine.

Primary objectives:

* To describe the persistence of anti-hepatitis B antibody at 9 to 10 years of age after last priming dose in subjects having received hepatitis B vaccine at birth and a hexavalent vaccine at 2, 4 and 6 months of age according to the vaccine received during A3L12 study (Hexaxim® [Group 1] or Infanrix® hexa [Group 2])
* To evaluate the immune response against hepatitis B one month after vaccination with a stand alone monovalent hepatitis B vaccine (challenge vaccination).

Secondary objectives:

* To describe serious adverse events (SAEs) reported throughout the trial after administration of hepatitis B vaccine.

DETAILED DESCRIPTION:
Subjects age 9 to 10 years who had received 3 injections of Hexaxim® or Infanrix® hexa and have completed the A3L12 study will be invited to participate in this study. They will receive one dose of Euvax-B® vaccine at Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by subject's parent/legally acceptable representative
* Assent form signed by subject
* Subject and parent(s)/legally acceptable representatives able to attend the scheduled visits and to comply with all trial procedures
* Receipt of primary vaccination with 3 doses of either Hexaxim® or Infanrix® hexa at the age of 2, 4, and 6 months in the A3L12 study, and hepatitis B vaccine at birth.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the inclusion in the trial
* Incomplete primary immunization in the A3L12 study
* Diagnostic of hepatitis B infection (clinical, serological, or virological confirmation) after completion of A3L12 study procedures
* Subjects known to have received hepatitis B vaccine after completion of the A3L12 study procedures
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination, except for Bacille Calmette Guerin (BCG) vaccination (any administration of oral polio vaccine [OPV] in the context of oral polio vaccine-national immunization days [OPV-NIDs] does not fall within the scope of this exclusion criterion)
* Receipt of any blood, blood-derived products or immunosuppressant drugs at the latest 3 months before inclusion
* Known or suspected diagnostic of congenital or acquired immunodeficiency since completion of the A3L12 study procedures
* Serious chronic illness occurring after receipt of the primary series (e.g., leukemia, lymphoma [T or B cells], Crohn's disease)
* Known or suspected subject seropositivity against human immunodeficiency virus (HIV) or hepatitis C since completion of the A3L12 study procedures
* Febrile (temperature ≥ 38.0°C) or acute, moderate or severe systemic illness on the day of inclusion.

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Levels of anti-Hepatitis B antibody concentrations in subject that received Hexaxim® or Infanrix® hexa vaccine in a previous study | Day 0 (pre-vaccination)
Levels of anti-Hepatitis B antibody concentrations in subject that received Hexaxim® or Infanrix® hexa vaccine in a previous study following vaccination with Euvax B® vaccine | Day 28 (post-vaccination)

SECONDARY OUTCOMES:
Number of subjects reporting Serious Adverse Events and relatedness to study vaccine throughout the study | Day 0 up to Day 28 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (2):
- Thailand (2):
  - Bangkok
  - Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com